CLINICAL TRIAL: NCT03769649
Title: Clinical Evaluation of Safety and Efficacy of the CelluTite Treatment
Brief Title: Clinical Evaluation of CelluTite Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO608110
Record Dates: First submitted 2018-12-04; First posted 2018-12-07 (Actual); Results first posted 2021-02-16 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2019-09

CONDITIONS: Cellulite of Thighs

STUDY DESIGN:
Intervention Model Description: Subjects will receive the treatment and outcome will be followed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment arm (Experimental): Subjects receive CelluTite treatment followed by Morpheus8 treatment
  Interventions: Device: CelluTite

INTERVENTIONS:
Device: CelluTite — CelluTite: Radiofrequency-assisted lipolysis (RFAL) Morpheus8: Fractional RF
  Other Names: Morpheus8

SUMMARY:
This prospective study is intended to evaluate the CelluTite RFAL handpiece combined with Morpheus8 handpiece for the treatment of cellulite.

DETAILED DESCRIPTION:
The study will evaluate the safety and efficacy of cellulite treatment using two hand pieces:

* The CelluTite - based on a minimally invasive, temperature-controlled Radiofrequency-assisted lipolysis (RFAL) technology. RF energy is applied using a handpiece with 2 electrodes: internal active electrode with spatula-shaped tip and external electrode.
* The Morpheus8 - designed to deliver RF energy to the skin surface in a fractional manner via an array of 24-electrode pins.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged 18-70 having mild/moderate grade cellulites.
* The patients should understand the information provided about the treatment, possible benefits and side effects, and sign the Informed Consent Form, (including the permission to use photography).
* The patients should be willing to comply with the study procedure and schedule, including the follow up visit, and will refrain from using any other aesthetic treatment methods in the treatment area for the last 6 months and during the entire study period.

Exclusion Criteria:

* Body fat layer thinner than 5mm.
* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body.
* Superficial permanent implant in the treated area such as metal plates and screws, metal piercing, silicone implants or an injected chemical substance.
* Current or history of skin cancer (remission of 5 years), or current condition of any other type of cancer, or pre-malignant moles.
* Severe concurrent conditions, such as cardiac disorders, epilepsy, uncontrolled hypertension, and liver or kidney diseases.
* Pregnancy and nursing.
* History of bleeding coagulopathies or use of anticoagulants.
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV or use of immunosuppressive medications.
* Poorly controlled endocrine disorders, such as diabetes or thyroid dysfunction and hormonal virilization.
* Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin.
* Use of Isotretinoin (Accutane®) within 6 months prior to treatment.
* Any surgery or treatment such as laser or chemicals in treated area within 3-6 months prior to treatment or before complete healing.
* Allergies, in particular to anesthesia.
* Mental disorders such as Body Dysmorphic Disorder (BDD).
* As per the practitioner's discretion, refrain from treating any condition that might make it unsafe for the patient.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Katz, MD, Principal Investigator — 60 E 56th St #2, New York, NY 10022, USA
Locations (1):
- Juva, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm
Started | 15
Completed | 11
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Population: Only subjects that finished all visits were analyzed
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.62 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 7
  Hispanic or Latino | 3
  Biracial | 1
Cellulite Score Rated According to Cellulite Severity Scale (Dimples) [Mean (Standard Deviation); unit: score on a scale] — Scale for evaluating cellulite dimples, in which a dimple is an isolated circular or oval-shaped depression on the surface of the skin. (A) Score 0 (no dimples); (B) score 1 (1 dimple); (C) score 2 (2 dimples); (D) score 3 (3 dimples); (E) score 4 (4 or more dimples). Higher values represent a worse outcome
  score on a scale | 3.45 (0.69)
Cellulite Score Rated According to Cellulite Severity Scale (Contour) [Mean (Standard Deviation); unit: score on a scale] — Scale for evaluating contour irregularities. The irregularities become more severe as more concavity and convexity occur in the linear undulations. Score 0-none-no depressions ; score 1 superficial: generalized, small depressions with no protuberances; score 2 mild: pattern of mild linear undulations; score 3 moderate: pattern of moderate linear undulations with alternating areas of protuberances and depressions; score 4 severe: severe generalized linear undulations with alternating areas of protuberances and depressions. higher values represent a worse outcome
  score on a scale | 3.55 (0.69)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cellulite Score Rated According to Cellulite Severity Scale (Dimples)
Description: Photos from 6 months follow-up visit will be evaluated. Evaluation goals are rating the degree of cellulite according to the Clinician Reported Photonumeric Cellulite Severity Scale (CR-PCSS). Scale for evaluating cellulite dimples, in which a dimple is an isolated circular or oval-shaped depression on the surface of the skin. (A) Score 0 (no dimples); (B) score 1 (1 dimple); (C) score 2 (2 dimples); (D) score 3 (3 dimples); (E) score 4 (4 or more dimples). Higher values represent a worse outcome
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
score on a scale | 2.45 (1.04)

2. Primary Outcome: Assessment of Occurrence of Adverse Events Based on Causality (Relationship to the Device or the Treatment)
Description: Safety will be evaluated by observation, assessment and recording of adverse events, if occur. Casualty: relationship to the device or the treatment 0 - no adverse event, 1 - not related and 2 - related to device). Higher values represent a worse outcome.
Time Frame: 6 months
Population: Only subjects completed 6 month FU
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Treatment Arm
Number analyzed (Participants) | 12
score | 0 (0)

3. Primary Outcome: Change in Cellulite Score Rated According to Cellulite Severity Scale (Contour)
Description: Photos from 6 months follow-up visit will be evaluated. Evaluation goals are rating the degree of cellulite according to the Clinician Reported Photonumeric Cellulite Severity Scale (CR-PCSS).
  Scale for evaluating contour irregularities. The irregularities become more severe as more concavity and convexity occur in the linear undulations. Score 0-none-no depressions ; score 1 superficial: generalized, small depressions with no protuberances; score 2 mild: pattern of mild linear undulations; score 3 moderate: pattern of moderate linear undulations with alternating areas of protuberances and depressions; score 4 severe: severe generalized linear undulations with alternating areas of protuberances and depressions. higher values represent a worse outcome
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
score on a scale | 2.64 (0.92)

4. Primary Outcome: Change in Cellulite Score Rated According to Cellulite Severity Scale (Contour)
Description: Photos from 1month follow-up visits will be evaluated. Evaluation goals are rating the degree of cellulite according to the Clinician Reported Photonumeric Cellulite Severity Scale (CR-PCSS).
  Scale for evaluating contour irregularities. The irregularities become more severe as more concavity and convexity occur in the linear undulations. Score 0-none-no depressions ; score 1 superficial: generalized, small depressions with no protuberances; score 2 mild: pattern of mild linear undulations; score 3 moderate: pattern of moderate linear undulations with alternating areas of protuberances and depressions; score 4 severe: severe generalized linear undulations with alternating areas of protuberances and depressions. higher values represent a worse outcome
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
score on a scale | 2.89 (0.93)

5. Primary Outcome: Change in Cellulite Score Rated According to Cellulite Severity Scale (Contour)
Description: Photos from 3 months follow-up visit will be evaluated. Evaluation goals are rating the degree of cellulite according to the Clinician Reported Photonumeric Cellulite Severity Scale (CR-PCSS). Scale for evaluating contour irregularities. The irregularities become more severe as more concavity and convexity occur in the linear undulations. Score 0-none-no depressions ; score 1 superficial: generalized, small depressions with no protuberances; score 2 mild: pattern of mild linear undulations; score 3 moderate: pattern of moderate linear undulations with alternating areas of protuberances and depressions; score 4 severe: severe generalized linear undulations with alternating areas of protuberances and depressions. higher values represent a worse outcome
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
score on a scale | 2.82 (0.87)

6. Primary Outcome: Change in Cellulite Score Rated According to Cellulite Severity Scale (Dimples)
Description: Photos 1 month follow-up visit will be evaluated. Evaluation goals are rating the degree of cellulite according to the Clinician Reported Photonumeric Cellulite Severity Scale (CR-PCSS). Scale for evaluating cellulite dimples, in which a dimple is an isolated circular or oval-shaped depression on the surface of the skin. (A) Score 0 (no dimples); (B) score 1 (1 dimple); (C) score 2 (2 dimples); (D) score 3 (3 dimples); (E) score 4 (4 or more dimples). Higher values represent a worse outcome
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
score on a scale | 2.6 (1.07)

7. Primary Outcome: Change in Cellulite Score Rated According to Cellulite Severity Scale (Dimples)
Description: Photos 3 month follow-up visit will be evaluated. Evaluation goals are rating the degree of cellulite according to the Clinician Reported Photonumeric Cellulite Severity Scale (CR-PCSS). Scale for evaluating cellulite dimples, in which a dimple is an isolated circular or oval-shaped depression on the surface of the skin. (A) Score 0 (no dimples); (B) score 1 (1 dimple); (C) score 2 (2 dimples); (D) score 3 (3 dimples); (E) score 4 (4 or more dimples). Higher values represent a worse outcome
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
score on a scale | 2.64 (0.81)

8. Primary Outcome: Change in Cellulite Score Rated According to Cellulite Severity Scale (Dimples)
Description: Photos 1 week follow-up visit will be evaluated. Evaluation goals are rating the degree of cellulite according to the Clinician Reported Photonumeric Cellulite Severity Scale (CR-PCSS). Scale for evaluating cellulite dimples, in which a dimple is an isolated circular or oval-shaped depression on the surface of the skin. (A) Score 0 (no dimples); (B) score 1 (1 dimple); (C) score 2 (2 dimples); (D) score 3 (3 dimples); (E) score 4 (4 or more dimples). Higher values represent a worse outcome
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
score on a scale | 1.9 (0.99)

9. Primary Outcome: Change in Cellulite Score Rated According to Cellulite Severity Scale (Contour)
Description: Photos from 1 week ollow-up visit will be evaluated. Evaluation goals are rating the degree of cellulite according to the Clinician Reported Photonumeric Cellulite Severity Scale (CR-PCSS). Scale for evaluating contour irregularities. The irregularities become more severe as more concavity and convexity occur in the linear undulations. Score 0-none-no depressions ; score 1 superficial: generalized, small depressions with no protuberances; score 2 mild: pattern of mild linear undulations; score 3 moderate: pattern of moderate linear undulations with alternating areas of protuberances and depressions; score 4 severe: severe generalized linear undulations with alternating areas of protuberances and depressions. higher values represent a worse outcome
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
score on a scale | 2 (0.82)

10. Primary Outcome: Assessment of Adverse Events Occurrence Based on Severity
Description: Safety will be evaluated by observation, assessment and recording of adverse events, if occur. Evaluations will be done based on severity (none 0, mild 1, moderate 2 or severe 3).
Time Frame: 3 months
Population: Only subjects completed 3 M FU were analyzed
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Treatment Arm
Number analyzed (Participants) | 12
score | 0 (0)

11. Primary Outcome: Assessment of Adverse Events Occurrence Based on Severity
Description: as for outcome 10
Time Frame: 1 month
Population: Only subjects completed 1 Month FU were analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 12
score on a scale | 0 (0)

12. Primary Outcome: Assessment of Adverse Events Occurrence Based on Severity
Description: as for outcome 10
Time Frame: 1 week
Population: Only subjects completed 1 week FU were analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 12
score on a scale | 0.08 (0.27)

13. Primary Outcome: Assessment of Adverse Events Occurrence Based on Severity
Description: as for outcome 10
Time Frame: Treatment Day
Population: All subjects undergone treatment were analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 15
score on a scale | 0.2 (0.41)

14. Primary Outcome: Assessment of Occurrence of Adverse Events Based on Causality (Relationship to the Device or the Treatment)
Description: as for outcome 2
Time Frame: 6 months
Population: Only subjects completed 6 months FU were analyzed
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
score | 0 (0)

15. Primary Outcome: Assessment of Adverse Events Occurrence Based on Severity
Description: as for outcome 10
Time Frame: 6 Months
Population: Only subjects completed 6 M FU were analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
score on a scale | 0 (0)

16. Primary Outcome: Assessment of Occurrence of Adverse Events Based on Causality (Relationship to the Device or the Treatment)
Description: as for outcome 2
Time Frame: 3 months
Population: Only subjects completed 6 months FU were analyzed
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Treatment Arm
Number analyzed (Participants) | 12
score | 0 (0)

17. Primary Outcome: Assessment of Occurrence of Adverse Events Based on Causality (Relationship to the Device or the Treatment)
Description: as for outcome 2
Time Frame: 1 week
Population: Only subjects completed 1 week FU were analyzed
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Treatment Arm
Number analyzed (Participants) | 12
score | 0.16 (0.55)

18. Primary Outcome: Assessment of Occurrence of Adverse Events Based on Causality (Relationship to the Device or the Treatment)
Description: as for outcome 2
Time Frame: Treatment Day
Population: Only subjects completed treatment were analyzed
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Treatment Arm
Number analyzed (Participants) | 15
score | 0.4 (0.8)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a period of 6 months
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 4/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=15)
Pain (Surgical and medical procedures) | 4 (4) — Anticipated event of pain post procedure in the treatment area that resolved after approximately a month.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT03769649/Prot_SAP_000.pdf